CLINICAL TRIAL: NCT04573894
Title: Diagnostic Performance of Plasma Procalcitonin in Screening for Contamination When Detecting Potential Contaminants in Blood Cultures
Brief Title: Diagnostic Performance of Plasma Procalcitonin for the Detection of Blood Cultures Contaminations
Status: Completed | Type: Observational
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Sponsor
Other Study IDs: 2020PI140
Record Dates: First submitted 2020-09-28; First posted 2020-10-05 (Actual); Last update posted 2020-10-05 (Actual); Status verified 2020-09

CONDITIONS: Blood Culture Contamination; Bacteremia; Contamination
Keywords: Procalcitonin
MeSH Terms: conditions — Bacteremia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — Positive blood cultures Procalcitonine
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Positives blood cultures: Collection of clinical and biological data of patients with blood cultures positives for potential contaminants, as well as PCT levels measurements, from January 2016 to May 2019 at the Nancy CHRU
  Interventions: Diagnostic Test: Procalcitonin dosage

INTERVENTIONS:
Diagnostic Test: Procalcitonin dosage — Plasma PCT levels measured by automated enzyme immunoassay (Kryptor).

SUMMARY:
In blood cultures, species considered as potentially contaminating (coagulase negative staphylococci (CNS), Bacillus spp., Corynebacterium spp., Cutibacterium acnes, Micrococcus spp., viridans group streptococci, and Clostridium perfringens) can, however, be responsable for true bacteremia.

Blood levels of the prohormone procalcitonin (PCT) markedly increase in the early stages of bacterial infections. The aim of our study is to determine the role of plasma PCT as a biomarker differentiating blood culture contaminations from true bacteremia.

DETAILED DESCRIPTION:
Blood culture contamination is defined by the introduction into of a microorganism into blood culture bottles from either the patient's or healthcare worker's flora, or the immediate environment during specimen collection. Species considered as potentially contaminating (coagulase negative staphylococci (CNS), Bacillus spp., Corynebacterium spp., Cutibacterium acnes, Micrococcus spp., viridans group streptococci, and Clostridium perfringens) can, however, be responsible for true bacteremia. If an organism belonging to one of those species is detected in isolates, rapidly and accurately assessing its contaminant or infectious potential is hence important to ensure effective antibiotic therapy as well as to reduce financial burden caused by unnecessary treatments, and additional clinical and laboratory costs.

Blood levels of the prohormone procalcitonin (PCT) markedly increase in the early stages of bacterial infections. The aim of our study is to determine the role of plasma PCT as a biomarker differentiating blood culture contaminations from true bacteremia.

ELIGIBILITY:
Inclusion Criteria:

* At least one blood culture positive for of the following microorganisms: coagulase negative staphylococci, viridans group streptococci
* PCT levels measurement on the day of blood culture specimen collection
* Adult patients

Exclusion Criteria:

* Patients with less than 3 blood culture bottles collected

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients hospitalized at the Nancy CHRU and at the Lorraine Cancer Institute (ICL) from January 2016 to May 2019 Patients screened for positive blood culture to one of the following microorganisms: coagulase negative staphylococci, viridans group streptococci; as well as procalcitonin levels measured at 24 hours.
Sampling Method: Non-Probability Sample
Enrollment: 147 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2020-07-31 (Actual); Study Completion 2020-09-05 (Actual)

PRIMARY OUTCOMES:
To evaluate the diagnostic potential of plasma procalcitonin in detecting blood culture contamination | 24 hours
  True contamination will be considered if all of the following biological criteria are met:
  * Only one bottle collected is positive
  * The growth time in the first positive bottle is more than 20 hours Plasma proclacitonin levels measured by automated enzyme immunoassay (Kryptor).

SECONDARY OUTCOMES:
To compare plasma PCT levels in patients with true bacteremia, probable bacteremia and contamination caused by the presence of bacterial species with high contaminant potential | 24 hours
  Bacteremia will be considered as present (" true bacteremia ") if all of the following biological criteria are met:
  * The same microorganism (amongst CNS, viridans group streptococci) is isolated in 100% of blood culture bottles collected from a given patient
  * The growth time in the first positive bottle is less than or equal to 16 hours
  Probable bacteremia:
  * When biological criteria of bacteremia and contamination are not fulled
  * When a antibiotic therapy is administrated without focal infection identified by cliniciens

CONTACTS AND LOCATIONS:
Locations (1):
- CHRU of Nancy, Nancy, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lu B, Shi L, Zhu F, Zhao H. Clinical Utility of the Time-to-Positivity/Procalcitonin Ratio to Predict Bloodstream Infection Due to Coagulase-Negative Staphylococci. Lab Med. 1 nov 2013;44(4):313-8.
- [Background] Schuetz P, Mueller B, Trampuz A. Serum procalcitonin for discrimination of blood contamination from bloodstream infection due to coagulase-negative staphylococci. Infection. 2007 Oct;35(5):352-5. doi: 10.1007/s15010-007-7065-0. Epub 2007 Sep 19. PMID 17882355
- [Background] Schuetz P, Albrich W, Mueller B. Procalcitonin for diagnosis of infection and guide to antibiotic decisions: past, present and future. BMC Med. 2011 Sep 22;9:107. doi: 10.1186/1741-7015-9-107. PMID 21936959
- [Derived] Berthezene C, Aissa N, Manteaux AE, Gueant JL, Oussalah A, Lozniewski A. Accuracy of procalcitonin for diagnosing peripheral blood culture contamination among patients with positive blood culture for potential contaminants. Infection. 2021 Dec;49(6):1249-1255. doi: 10.1007/s15010-021-01697-4. Epub 2021 Sep 15. PMID 34524647